CLINICAL TRIAL: NCT01534052
Title: A Phase 2 Open-label Extension Study to Assess the Safety of Continued Administration of MDV3100 in Subjects With Prostate Cancer Who Showed Benefit From Prior Exposure to MDV3100
Brief Title: A Study to Assess the Safety of Continued Administration of MDV3100 in Subjects With Prostate Cancer Who Showed Benefit From Prior Exposure to MDV3100
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9785-CL-0121
Record Dates: First submitted 2012-02-08; First posted 2012-02-16 (Estimated); Results first posted 2018-04-27 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Castration-Resistant Prostate Cancer (CRPC)
Keywords: Prostate Cancer; Castration-Resistant Prostate Cancer (CRPC); MDV3100; Androgen receptor signaling inhibitor
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Enzalutamide (Experimental): Participants received 160 mg enzalutamide orally once a day. Participants continued on treatment unless the dose was reduced or treatment was interrupted during the study.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — Oral
  Other Names: MDV3100; ASP9785; Xtandi

SUMMARY:
A study to assess the safety of continued administration of MDV3100 in subjects with Prostate Cancer who have already undergone treatment with MDV3100 and showed benefit.

DETAILED DESCRIPTION:
This was a multi-center extension study in participants with prostate cancer who have completed MDV3100 treatment study to assess the long-term safety of continued administration of MDV3100, when judged by the investigator to be in the best interest of the participant. For the study duration, all participants with castration-resistant prostate cancer (CRPC) maintained androgen deprivation with a Luteinizing Hormone Releasing Hormone (LHRH) agonist/antagonist unless they underwent bilateral orchiectomy. Participants were discontinued from study drug when the continued administration of study drug was deemed to be not in the participants' best interest by the investigator based on clinical assessment. Throughout the study, safety and tolerability were assessed by the recording of adverse events, monitoring of vital signs and physical examinations, safety laboratory evaluations, and 12-lead electrocardiograms (ECGs). Participants had a safety follow-up visit 30 days after their last dose of study drug. Participants that did not meet any of the discontinuation criteria were eligible to continue to receive treatment with enzalutamide in study 9785-CL-0123 [NCT02960022] upon approval and activation of the study at the participating institution. Participants who enrolled in study 9785-CL-0123 [NCT02960022] were not required to have a safety follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Has completed a prior study with MDV3100, can be enrolled in this extension study without any interruption in study drug
* No new clinically significant abnormalities based upon physical examination, safety laboratory data, vital signs, ECG, and other clinical assessments noted from the last visit conducted during the subject's active MDV3100 study prior to initiation of this study
* Male subjects and their female spouses/partners who are of childbearing potential must be using highly effective contraception1 consisting of two forms of birth control (one of which must be a barrier method) starting at Screening and continue throughout the study period and for 3 months after final study drug administration. Male subjects must not donate sperm starting at Screening and throughout the study period and for at least 3 months after final study drug administration. 1Highly effective contraception is defined as:

  * Established use of oral, injected or implanted hormonal methods of contraception.
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS).
  * Barrier methods of contraception: Condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal form/gel/film/ cream/suppository
* Subject agrees not to participate in another interventional study while on treatment

Exclusion Criteria:

Subject will be excluded from participation if any of the following apply:

1. Subject has a history of seizure or any condition that may predispose to seizure including, but not limited to underlying brain injury, stroke, primary brain tumours, brain metastases, or alcoholism.
2. Subject has a history of loss of consciousness or transient ischemic attack within 12 months prior to Day 1 of the completed preceding study.
3. Use of the following prohibited medication/therapies:

   * Concomitant medication that likely could cause clinically relevant drug-to-drug interactions with MDV3100.
   * Other (than MDV3100) androgen-receptor (AR) antagonists (bicalutamide, flutamide, nilutamide).
   * Investigational therapy other than MDV3100 or investigational procedures of any kind.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-10-21 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (7):
- United States (4):
  - Site US107, Aurora, Colorado
  - Site US104, Chicago, Illinois
  - Site US105, Pittsburgh, Pennsylvania
  - Site US106, San Antonio, Texas
- Site MD37301, Chisinau, Moldova
- South Africa (2):
  - Site ZA2701, George
  - Site ZA2702, Port Elizabeth

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=241

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 1 site in the Republic of Moldova, 2 sites in South Africa and 4 sites in the United States. In order to participate, participants had to complete a prior study with enzalutamide, be in a state of at least stable disease and benefit from continued treatment with enzalutamide in the opinion of the investigator.
Pre-assignment Details: This was an extension study in prostate cancer participants who have received enzalutamide treatment in prior phase 1 studies. The 9785-CL-0121 was an extension of previous enzalutamide studies (9785-CL-0003 [NCT01902251], 9785-CL-0007 [NCT01911728] & 9785-CL-0406 [NCT02225093]).
Period: Overall Study
Arm/Group | Enzalutamide
Started | 52
Treatment Received | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The analysis population was the Safety Analysis Set (SAF), which consisted of participants who received at least one dose of enzalutamide during the extension study. This extension study's baseline was considered the original baseline from the prior parent studies with enzalutamide.
Arm/Group | Enzalutamide
Number analyzed (Participants) | 52
Age, Continuous [Geometric Mean (Standard Deviation); unit: years] | 68.6 (7.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 47
  More than one race | 0
  Unknown or Not Reported | 3
Duration of Prostate Cancer [Geometric Mean (Standard Deviation); unit: months] — The duration of prostate cancer was calculated as (Date of first enzalutamide intake in the parent study - Date of initial diagnosis) + 1.
  months | 69.4 (64.10)
Primary Gleason Score at Initial Diagnosis [Count of Participants; unit: Participants] — Gleason score was a grading system for prostate cancer tissue based on how it looks under a microscope. Gleason scores ranged from 2 to 10 and indicated how likely it was that a tumor will spread. A low Gleason score meant the cancer tissue is similar to normal prostate tissue and the tumor was less likely to spread; a high Gleason score meant the cancer tissue was very different from normal and the tumor was more likely to spread.
  Participants
    Score 3 | 15
    Score 4 | 13
    Score 5 | 4
    Unknown | 20
Secondary Gleason Score at Initial Diagnosis [Count of Participants; unit: Participants] — Gleason score was a grading system for prostate cancer tissue based on how it looks under a microscope. Gleason scores ranged from 2 to 10 and indicated how likely it was that a tumor will spread. A low Gleason score meant the cancer tissue is similar to normal prostate tissue and the tumor was less likely to spread; a high Gleason score meant the cancer tissue was very different from normal and the tumor was more likely to spread.
  Participants
    Score 3 | 9
    Score 4 | 14
    Score 5 | 9
    Unknown | 20
Total Gleason Score at Initial Diagnosis [Count of Participants; unit: Participants] — Gleason score was a grading system for prostate cancer tissue based on how it looks under a microscope. Gleason scores ranged from 2 to 10 and indicated how likely it was that a tumor will spread. A low Gleason score meant the cancer tissue is similar to normal prostate tissue and the tumor was less likely to spread; a high Gleason score meant the cancer tissue was very different from normal and the tumor was more likely to spread.
  Participants
    Score 6 | 5
    Score 7 | 16
    Score 8 | 1
    Score 9 | 13
    Unknown | 17
Primary Tumor Assessment at Initial Diagnosis - Clinical Tumor Stage (T) [Count of Participants; unit: Participants]
  TX - Primary Tumor Cannot be Assessed | 3
  T0 - No Evidence of Primary Tumor | 1
  T1 - Clinically Tumor Not Palpable or Visible | 1
  T2 - Tumor Confined Within the Prostate | 8
  T3 - Tumor Extends Through the Prostatic Capsule | 13
  T4 - Tumor Fixed or Invades Adjacent Structures | 3
  Unknown | 23
Pathologic Tumor Stage (pT) [Count of Participants; unit: Participants]
  pT2 - Organ Confined | 5
  pT3 - Extraprostatic Extension | 9
  pT4 - Invasion of Bladder, Rectum | 1
  Unknown | 37
Regional Lymph Nodes (N) at Initial Diagnosis [Count of Participants; unit: Participants]
  NX - Regional Lymph Nodes Were Not Assessed | 18
  N0 - No Regional Lymph Node Metastasis | 15
  N1 - Metastasis in Regional Lymph Node(s) | 6
  pNX - Regional Lymph Nodes Not Sampled | 8
  pN0 - No Positive Regional Nodes | 6
  pN1 - Metastasis in Regional Nodes(s) | 2
  Unknown | 36
Distant Metastasis at Initial Diagnosis [Count of Participants; unit: Participants]
  MX - Distant Metastasis Cannot be Assessed | 8
  M0 - No Distant Metastasis | 12
  M1 - Distant Metastasis | 9
  Unknown | 23
Treatment Duration in Extension Study [Number; unit: Days] — Treatment duration in the extension study was calculated as (Date of last dose of MDV3100 - Date of first dose of MDV3100 in the extension study)+ 1.
  Days
    <= 60 | 4
    > 60 - <182 | 12
    >= 182 - <365 | 9
    >= 365 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered study drug or who underwent study procedures and did not necessarily have a causal relationship with treatment. An abnormality identified during a medical test was defined as an AE only if the abnormality induced clinical signs or symptoms, required active intervention, required interruption, or discontinuation of study medication, or was clinically significant in the opinion of the investigator. An AE was defined as serious if it resulted in any of the following outcomes: Death, Was life-threatening, Persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, Congenital anomaly, or birth defect, Inpatient hospitalization or prolongation of hospitalization, Other medically important event. Drug-related AEs were those assessed by the investigator as AEs whose relationship to the to the study drugs could not be ruled out.
Time Frame: From the date of the first dose of study drug to 30 days after last dose of study drug; the median duration of treatment was 392 days, and the maximum was 1926 days
Population: The analysis population was the SAF.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 52
Participants
  Any TEAE | 43
  Drug-Related TEAEs | 27
  Deaths | 5
  Serious TEAEs | 17
  Drug-Related Serious TEAEs | 5
  TEAEs Leading to Study Drug Discontinuation | 12
  Drug-Related TEAEs Lead to Study Discontinuation | 5

ADVERSE EVENTS:
Time Frame: From the date of the first dose of study drug to 30 days after last dose of study drug; the median duration of treatment was 392 days, and the maximum was 1926 days
Description: The total number of deaths (all causes) includes deaths reported after the time frame above.
Groups:
- Enzalutimide: Participants received 160 mg enzalutamide orally once a day. Participants continued on treatment unless the dose was reduced or treatment was interrupted during the study.
Arm/Group | Enzalutimide
All-Cause Mortality (participants affected / at risk) | 2/52
Serious Adverse Events (participants affected / at risk) | 17/52
Other Adverse Events (participants affected / at risk) | 33/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutimide (N=52)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutimide (N=52)
Anaemia (Blood and lymphatic system disorders) | 4 (6)
Constipation (Gastrointestinal disorders) | 5 (7)
Diarrhoea (Gastrointestinal disorders) | 5 (8)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (4)
Fatigue (General disorders) | 14 (21)
Weight decreased (Investigations) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (4)
Pollakiuria (Renal and urinary disorders) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 3 (3)
Hot flush (Vascular disorders) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. The sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2016-06-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT01534052/Prot_000.pdf
  • Statistical Analysis Plan (2015-04-08): https://cdn.clinicaltrials.gov/large-docs/52/NCT01534052/SAP_001.pdf